CLINICAL TRIAL: NCT03874000
Title: An Open-Label Single-Arm Phase Ⅱ Study to Evaluate Efficacy and Safety of Sintilimab Combined With Metformin Hydrochloride in Patients With Advanced Non-small Cell Lung Cancer Refractory to First-Line Treatment
Brief Title: Sintilimab Combined With Metformin in First-Line Chemotherapy Refractory Advanced NSCLC Patients
Acronym: SMART
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMART
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2018-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Sintilimab; Metformin Hydrochloride; second line; cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — sintilimab; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab plus Metformin Hydrochloride (Experimental): Patients receive metformin hydrochloride 500mg orally (PO) twice daily (BID). Patients also receive Sintilimab 200mg intravenously (IV) in 60 minutes on day 1. Courses repeat every 21 days in the absence of disease progression, unacceptable toxicity, or withdrawal of consent.
  Interventions: Biological: Sintilimab; Drug: Metformin Hydrochloride

INTERVENTIONS:
Biological: Sintilimab — Given IV
  Other Names: IBI308
Drug: Metformin Hydrochloride — Given PO
  Other Names: Glucophage

SUMMARY:
Evaluate the Efficacy and Safety of Sintilimab Combined with Metformin Hydrochloride in Patients with Advanced Non-small Cell Lung Cancer Refractory to First-Line Platinum-Containing Chemotherapy

DETAILED DESCRIPTION:
This study is an open-label, single-arm, phase II clinical study on the efficacy and safety of Sintilimab combined with metformin in the treatment of locally advanced, recurrent or metastatic NSCLC patients who fail to receive first-line platinum-containing chemotherapy in patients with locally advanced, recurrent or metastatic non-small-cell lung cancer in China. Simon two stages optimal design criteria are used in the test, and 18 subjects are enrolled in the first stage, and if two or more patients reach the PR/CR evaluation criteria, the sample size will be increased to 43. If 7 or more of the 43 subjects meets the PR/CR evaluation criteria, it indicates that the test achieves the expected results. After the subject signs the informed consent, the subject will receive the treatment of 200 mg IV Q3W (3 weeks using a) of Sintilimab combine with 500mg of metformin for oral bid until disease progression, death, toxicity intolerance, withdrawal of the informed consent, initiation of new anti-tumor treatment or termination of treatment for other reasons specified in the program. The longest duration of treatment for Sintilimab is 24 months. The main endpoint of the study is ORR evaluated by the researchers based on RECIST v1.1.

RECIST v1.1 is used for clinical tumor imaging evaluation. Based on the clinical conditions of the patients, it is used every 2 cycles (±7 days) until disease progression, initiation of new anti-tumor therapy, withdrawal of Inform Consent Form (ICF) or death of the subjects. For the first time, if the clinical status of the subjects with disease progression is stable, those who meet the criteria determined by the investigator can continue to receive treatment of Sintilimab combined with metformin, and must undergo imaging evaluation after 4 weeks (± 7 days) to confirm the disease progression. Patients with disease progression will enter the survival follow-up stage (every 60 ± 7 days); Patients who stop treatment due to other causes other than disease progression will continue to receive the tumor assessment every 6 weeks (± 7 days) until the next event (initiation of new anti-tumor treatment, disease progression, withdrawal of ICF or death), and then enter the survival follow-up stage (every 60 ± 7 days).

The investigator will evaluate and manage the adverse reactions during the treatment period and within 30 ± 7 days after the last use of the study drug in accordance with the NCI Common Terminology Criteria for Adverse Events (CTCAE) 4.0 and immune-related adverse reactions standard Immune-Related Response Criteria (irRC), evaluation and management of severe adverse reactions during the treatment period and 90 ± 7 days after the last use of the study drug (unless patients start new anti-tumor treatment 31 to 90 days after the last use of the study drug).

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent forms
2. Male or female,18-75 years of ages
3. Eastern Cooperative Oncology Group (ECOG) PS：0-2
4. Life expectancy of more than 12 weeks
5. Histologically or cytologically confirmed, non-small cell lung cancer (NSCLC) (the participant who has undergone pathological re-examination asked to take the site that had not received radiotherapy)
6. Locally advanced, metastatic or recurrent [unresectable or not meet the standard of radical radiotherapy and chemotherapy IIIB, IIIC or IV NSCLC, according to the 8th Edition of the Union Internationale Contre le Cancer (UICC)/American Joint Committee on Cancer (AJCC) Staging system] NSCLC
7. Both cases are received by first-line platinum chemotherapy failed

1). First-line platinum chemotherapy during or after treatment (include maintenance treatment) are defined by initial progressive disease (PD) (RECIST v1.1), during first-line platinum chemotherapy received one drug was discontinued, reduced or replaced with a similar drug 2). For recurrent disease≤6 months, adjuvant chemotherapy, neoadjuvant chemotherapy or neoadjuvant chemotherapy plus adjuvant chemotherapy may be accepted, participants must have histologically confirmed, not epidermal growth factor receptor (EGFR) mutation or anaplastic lymphoma kinase (ALK) translocation 8. Histologically confirmed participants without EGFR mutation or ALK/c-ros oncogene 1 receptor kinase (ROS1) rearrangement 9. At baseline, subjects will be required to provide fresh tissue biopsy specimens, and biopsy specimens should be confirmed by a pathologist 10. Participants must have a measurable disease (RECIST v1.1) 11. At baseline, glycated hemoglobin (HbA1C)≤6.4% 12. Important organs and bone marrow functions meet the following requirements (All tests should be completed two weeks before medication, expect the participants treated with any cell and growth factor within two weeks)

1. . Blood routine: Absolute neutrophil (ANC)≥1.5×109/L, platelets (PLT)≥10×109/L, Hemoglobin (HGB)≥90g/L, (No transfusion or erythropoietin dependence≤14days)
2. . Liver functions: Total bilirubin ≤1.5 times the institutional upper limit of normal (ULN), Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SPGT])≤2.5 X institutional ULN (or≤5 times ULN in case of liver metastasis)
3. . Renal functions: Creatinine(Cr)≤1.5×ULN,or creatinine clearance (CrCl)≥60milliliter (mL)/min (use Cockcroft-Gault formula) Female: CrCl=(140-age) ×weight(kg) ×0.85/72×Cr(mg/dL) Male: CrCl=(140-age) ×weight(kg) ×1.00/72×Cr(mg/dL) 13. Coagulation function: international normalized ratio(INR) or prothrombin time (PT)≤1.5 ULN; If the subject is receiving anticoagulant treatment, INR will be sufficient as long as the anticoagulant is within the prescribed range of use 14. No brain metastasis was confirmed by plain scanning and enhanced MRI /CT examination within 2 weeks before medication; Asymptomatic brain metastasis, or symptomatic brain metastasis participants who have received stereotactic radiosurgery (SRS) or whole-brain radiation therapy (WBRT) in the past, may also be included in the test if the lesion is not enlarged or the central nervous system symptoms are not evaluated by cranial MRI within 4 weeks before enrollment 15. For women of child-bearing age, a negative urine or serum pregnancy test should be conducted 3 days prior to the first study drug administration 16. Subject and subject's sexual partner will be required to use a medically approved contraceptive (such as an intrauterine device, contraceptive or condom, etc.) during and within 6 months after the study treatment period

Exclusion Criteria:

1. Participants should not have received metformin within 6 months prior to registration
2. In the past, participants have received anti PD-1, anti PD-L1 or anti PD-L2 drugs or drugs targeting another stimulation or synergistic inhibition of T cell receptors (such as Cytotoxic T-Lymphocyte Antigen 4 [CTLA-4] and CD137)
3. Received the following treatment:

   Within 2 weeks before the first administration, 1). Received systemic therapy with Chinese adult drugs or immunomodulatory drugs (including thymosine and interferon, except for topical use to control pleural effusion) with anticancer indications 2). 4 weeks prior to the first administration, received any investigational drug therapy or use of research instruments 3). Receive an overdose of immunosuppressive agents (systemic glucocorticoid over 10 mg/ day prednisone or its equivalent) within 4 weeks prior to the first dose 4). Live vaccine was given within 4 weeks before the first dose Note: inactivated virus vaccine for seasonal influenza is allowed within 30 days prior to the first dose, but live attenuated influenza vaccine for intranasal administration is not allowed 5). Major surgery (such as an open cavity, thoracotomy, or laparotomy), or unhealed surgical wounds, ulcers, or fractures, has been performed within 4 weeks prior to the first administration 6). The adverse reactions of any previous anti-tumor treatment did not return to CTCAE ≤level 1(excluding hair loss and laboratory tests without clinical significance).
4. Participants who suffer from type 1 or type 2 diabetes, or high blood sugar that require medication
5. Active autoimmune diseases requiring systemic therapy (e.g. the use of disease-relieving drugs/corticosteroids or immunosuppressants) occurred within 2 years prior to the first administration. Alternative therapies (such as thyroxine or physiological corticosteroids for adrenal or pituitary insufficiency) are not considered systemic
6. Allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation are known
7. Allergic reaction to the active ingredients or any adjuncts of Sintilimab or metformin
8. History of lactic acid or other metabolic acidosis
9. Symptomatic central nervous metastasis and/or cancerous meningitis
10. Interstitial pulmonary disease or previous lung disease requires oral or intravenous hormone control
11. Clinically uncontrollable third interstitial effusion, such as pleural and ascites, which cannot be controlled by drainage or other methods before enrollment
12. Other malignancies were diagnosed within 5 years prior to the first administration, with the exception of radical cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, and/or radical carcinoma in situ
13. Suffering from other serious uncontrollable diseases, including but not limited to 1). Kidney disease or renal dysfunction caused by heart failure (shock), acute myocardial infarction, sepsis, etc. [serum creatinine(Cr)≥1.5mg/dL (male), ≥ 1.4mg/dL (female) or creatinine clearance rate (CrCl)≤ 60mL/min] 2). Congestive heart failure requiring medication (grade III to IV, New York Heart Association [NYHA] classification), unstable angina, poorly controlled and clinically significant arrhythmia 3). A severe infection that requires medical treatment 4). Past cardiopulmonary disease, current need drugs or oxygen support 5). Chronic alcoholism or risk of chronic alcoholism was assessed by investigator 6). HIV Infected person (HIV antibody positive) 7). Untreated active hepatitis b Note: Subjects with hepatitis b who meet the following criteria are also eligible for inclusion: before the first dose, hepatitis B virus (HBV) DNA is less than 1×103 copy number /ml (200IU/ ml), and subjects should receive anti-HBV treatment throughout the study to avoid reactivation of the virus 8). For subjects with anti-hepatitis B core antigen (HBC) (+), HBsAg (-), anti-HBs (-), and HBV viral load (-), prophylactic anti-HBV therapy is not required, but virus reactivation is monitored closely 9). Subjects with active HCV infection (HCV antibody positive and HCV-RNA level higher than the detection limit) 10). Active tuberculosis, etc 11). Any arterial thrombosis, embolism or ischemia, such as cerebrovascular accident or transient ischemic attack, occurred within 6 months before the inclusion of treatment 12). Clinical active diverticulitis, abdominal abscess, gastrointestinal ulcer, etc 13). Uncontrolled hypercalcemia (> 1.5 mmol/L of calcium ions or > 12 mg/dL of calcium or serum calcium > ULN after correction) or symptomatic hypercalcemia requiring continued bisphosphonate therapy
14. Other acute or chronic disease, mental illness, or laboratory abnormalities that may result in increased risk of study participation or drug administration, or interfere with the interpretation of the study results, and disqualify participants from participating in the study according to the judgment of the investigator
15. Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2019-03-08 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-06-05 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  ORR is defined as participants who had complete response (CR) or partial response(PR) divided by the total number of patients.

SECONDARY OUTCOMES:
Overall Survival (OS) | From enrollment until death (up to 24 months)
  OS is defined as time from date of enrollment to date of death due to any cause. For participants still alive at the time of analysis, OS time was censored on last date that participants were known to be alive.
Progress free survival (PFS） | each 42 days up to PD or death (up to 24 months)
  The PFS time is defined as time from enrollment to locoregional or systemic recurrence, second malignancy or death due to any cause; censored observations will be the last date of : "death", "last tumor assessment", "last follow up date" or "last date in drug log"
Disease Control Rate (DCR） | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  DCR is defined as the percentage of participants with Disease Control best overall response (complete response, partial response or stable disease).
Duration of Response (DOR) | From the first response date to PD or death (up to 24 months)
  For participants with response (CR or PR), the duration of response: the time from the first response date to disease progression or death, and the date of the final imaging evaluation was deleted for participants without PD or death.

CONTACTS AND LOCATIONS:
Overall Officials: Dingzhi Huang, M.D., Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access requests will be reviewed by an external independent Review Panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Result] Kubo T, Ninomiya T, Hotta K, Kozuki T, Toyooka S, Okada H, Fujiwara T, Udono H, Kiura K. Study Protocol: Phase-Ib Trial of Nivolumab Combined With Metformin for Refractory/Recurrent Solid Tumors. Clin Lung Cancer. 2018 Nov;19(6):e861-e864. doi: 10.1016/j.cllc.2018.07.010. Epub 2018 Aug 9. PMID 30172698
- [Result] Afzal MZ, Mercado RR, Shirai K. Efficacy of metformin in combination with immune checkpoint inhibitors (anti-PD-1/anti-CTLA-4) in metastatic malignant melanoma. J Immunother Cancer. 2018 Jul 2;6(1):64. doi: 10.1186/s40425-018-0375-1. PMID 29966520